CLINICAL TRIAL: NCT00302250
Title: Study of The Effect of Vascular Distensibility on Endothelial-Dependent Vasoreactivity in Subjects With Systolic Hypertension Before and After Receiving Oral Alagebrium or Placebo for 8 Weeks (STRETCH)
Brief Title: The STRETCH Study: Distensibility on Endothelial-Dependent Vasoreactivity in Subjects With Systolic Hypertension
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Synvista Therapeutics, Inc (Industry)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart and Lung Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ALT-711-0217 (Amended)
Record Dates: First submitted 2006-03-13; First posted 2006-03-14 (Estimated); Last update posted 2006-03-22 (Estimated); Status verified 2006-03

CONDITIONS: Cardiovascular Disease
Keywords: Cardiovascular; Flow-mediated vasodilation (FMD); Pulse perfusion-mediated vasodilation (PPMV); Endothelial function; Heart failure
MeSH Terms: conditions — Cardiovascular Diseases; Heart Failure | interventions — alagebrium

INTERVENTIONS:
Drug: ALT-711 (alagebrium chloride)

SUMMARY:
The primary objective of the double-blind segment is to compare effects of alagebrium vs placebo on change from baseline in endothelial function, as assessed by flow-mediated vasodilation (FMD).

DETAILED DESCRIPTION:
The secondary objectives of the double-blind segment are to:

* Compare the effects of alagebrium vs placebo on the change from baseline in endothelial-mediated vasoreactivity immediately after exercise, as assessed by pulse perfusion-mediated vasodilation (PPMV).
* Confirm results observed in the single-blind segment.
* Explore several variables as potential independent predictors of vascular stiffness and endothelial function. These parameters include age, body mass index, gender, renal disease, history of cardiovascular disease, serum cholesterol, and antihypertensive medication use.
* Provide insight into nitric oxide-dependent endothelial function in the setting of increased arterial stiffness by determination of substances in the nitric oxide signaling pathway (specifically, levels of serum cGMP; serum nitrate and nitrite; and serum asymmetric dimethylarginine [ADMA], an endogenous inhibitor of nitric oxide synthase).
* Provide insight into the relationship between AGE levels (AGE markers: pentosidine, furosine), collagen metabolism (collagen markers: procollagen I carboxyterminal propeptide [PICP], procollagen type I N terminal propeptide [PINP], cross-linked carboxyterminal telopeptide of Type I collagen [ICTP], n-terminal propeptide of type III procollagen [PIIINP]), and endothelial function; and insight into the changes in these markers in response to treatment with an AGE cross-link breaker (alagebrium).
* Provide insight into the relationship between markers of inflammation [specifically, free and total serum matrix metalloproteinase-1(MMP-1), free tissue inhibitor of metalloproteinase 1 (TIMP1), intercellular adhesion molecule-1 (ICAM), vascular cellular adhesion molecule (VCAM), P-selectin, von Willebrand factor (vWf), interleukin-6 (IL-6), endothelin 1, VEGF, NFkβ, TGF-β, IGF-1 and high-sensitivity C reactive protein (hs CRP)] and endothelial function; and insight into the changes in these markers in response to treatment with an AGE cross-link breaker (alagebrium).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female 50 years of age or greater.
2. Diagnosed with systolic hypertension (systolic blood pressure >140 mm Hg and (less than or equal to) 200 mm Hg, and a diastolic blood pressure (less than or equal to) 95 mm Hg) and elevated pulse pressure (systolic blood pressure [SBP] minus diastolic blood pressure [DBP] greater than 60 mm Hg).
3. Normal left ventricular function (ejection fraction > 55%) at baseline (Visit 3).
4. Brachial artery must be able to be visualized for FMD and PPMV determinations.
5. Able to perform bicycle exercise.
6. Able to read, understand and sign the informed consent after the nature of the study has been explained.
7. If sexually active, the subject agrees to use reliable contraception while participating in this study. If a woman, is surgically sterilized or post-menopausal, or has a negative serum pregnancy test.

Exclusion Criteria:

1. Aortic stenosis, prior known coronary artery disease (including myocardial infarction), cerebrovascular accident, or peripheral vascular disease.
2. Uncontrolled hypertension (SBP > 200/DBP > 95 mm Hg).
3. Atrial fibrillation, diabetes mellitus treated with insulin, or chronic lung disease.
4. Any additional condition(s) which, in the opinion of the investigator, would prohibit the subject from completing the study, or not be in the best interest of the subject.
5. Treatment with nitrates, or a change in antihypertensive medications within the last 1 month.
6. Treatment with any investigational drug within 1 month prior to study drug administration.
7. Previous exposure to alagebrium.
8. AST (SGOT) or ALT (SGPT) > 2x normal limit.
9. Serum creatinine > 2.0 mg/dL.
10. Cigar/cigarette smoking.
11. Necessity to use smokeless tobacco or nicotine-containing products, or to consume caffeine, alcohol, or antioxidants starting at midnight prior to study clinic visits. NOTE: Water is allowed ad libitim.
12. Positive drug screen.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70
Dates: Start 2006-02; Study Completion 2006-12

CONTACTS AND LOCATIONS:
Overall Officials: Susan Zieman, MD, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University School of Medicine, Baltimore, Maryland, United States

REFERENCES:
- [Background] Little WC, Zile MR, Kitzman DW, Hundley WG, O'Brien TX, Degroof RC. The effect of alagebrium chloride (ALT-711), a novel glucose cross-link breaker, in the treatment of elderly patients with diastolic heart failure. J Card Fail. 2005 Apr;11(3):191-5. doi: 10.1016/j.cardfail.2004.09.010. PMID 15812746
- [Background] Kass DA, Shapiro EP, Kawaguchi M, Capriotti AR, Scuteri A, deGroof RC, Lakatta EG. Improved arterial compliance by a novel advanced glycation end-product crosslink breaker. Circulation. 2001 Sep 25;104(13):1464-70. doi: 10.1161/hc3801.097806. PMID 11571237
- [Background] Liu ZR, Ting CT, Zhu SX, Yin FC. Aortic compliance in human hypertension. Hypertension. 1989 Aug;14(2):129-36. doi: 10.1161/01.hyp.14.2.129. PMID 2759675
- [Background] Corretti MC, Anderson TJ, Benjamin EJ, Celermajer D, Charbonneau F, Creager MA, Deanfield J, Drexler H, Gerhard-Herman M, Herrington D, Vallance P, Vita J, Vogel R; International Brachial Artery Reactivity Task Force. Guidelines for the ultrasound assessment of endothelial-dependent flow-mediated vasodilation of the brachial artery: a report of the International Brachial Artery Reactivity Task Force. J Am Coll Cardiol. 2002 Jan 16;39(2):257-65. doi: 10.1016/s0735-1097(01)01746-6. PMID 11788217